CLINICAL TRIAL: NCT02825875
Title: Study of the Clinical Utility of PSMA Imaging in the Evaluation of Men With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: J15216; IRB00084971 (Other: JHM IRB)
Record Dates: First submitted 2016-06-30; First posted 2016-07-07 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adenocarcinoma of the prostate
  Interventions: Drug: 18F DCFPyL- Radiopharmaceutica

INTERVENTIONS:
Drug: 18F DCFPyL- Radiopharmaceutica

SUMMARY:
In this study we aim to more precisely define the clinical utility of PSMA imaging across a range of clinical indications in men with prostate cancer. To accomplish this, we will make the 18F-DCFPyL PET/CT scan available to urologists, medical oncologists, and radiation oncologists at Johns Hopkins and survey physicians as to the indication for ordering the PET/CT and if a change in management occurred as the result of new information gained from the scan. We believe these data will prove critical for planning future studies aimed at evaluating the efficacy of this test for improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Willingness to signed informed consent
3. Histologically confirmed adenocarcinoma of the prostate
4. PSA measurement ≤60 days prior to study enrollment
5. Completed radiographic evaluation with whole-body bone scan (99mTc-MDP or Na18F) and cross-sectional imaging (CT or MRI) of the abdomen and pelvis ≤60 days prior to study enrollment

Exclusion Criteria:

1. Administered a radioisotope within 5 physical half-lives prior to study enrollment
2. History of other malignancy diagnosed within the last 5 years (exceptions: low grade urothelial carcinoma of the bladder, squamous cell carcinoma or basal cell carcinoma of the skin).

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adenocarcinoma of the prostate
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Physician responses to a questionnaire | less than 1 year
  The Post-PET/CT questionnaire will determine if the PET/CT scan results in changes to clinical management of patient illness.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gorin, MD, Principal Investigator — Professor of Oncology
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States